CLINICAL TRIAL: NCT00744926
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Effect of Taspoglutide Compared to Placebo, in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Diet and Exercise
Brief Title: A Study of Taspoglutide Versus Placebo for the Treatment of Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Diet and Exercise.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC20750; 2008-001765-28
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- taspoglutide 10mg sc (Experimental)
  Interventions: Drug: taspoglutide
- taspoglutide 10mg/20mg sc (Experimental)
  Interventions: Drug: taspoglutide

INTERVENTIONS:
Drug: placebo — sc, once weekly
  Arms: placebo
Drug: taspoglutide — 10mg sc, once weekly
  Arms: taspoglutide 10mg sc
Drug: taspoglutide — 20mg sc, once weekly (after 4 weeks of taspoglutide 10mg sc once weekly)
  Arms: taspoglutide 10mg/20mg sc

SUMMARY:
This 3 arm study will assess the efficacy, safety and tolerability of taspoglutide compared to placebo in patients with type 2 diabetes mellitus inadequately controlled with diet and exercise. Patients will be randomized to one of 3 treatment arms: taspoglutide 10mg sc once weekly, taspoglutide 20mg sc once weekly (after 4 weeks of taspoglutide 10mg sc once weekly) or placebo. After the first 24 weeks patients on placebo will be switched to taspoglutide 10mg once weekly or taspoglutide 20mg once weekly (after 4 weeks of taspoglutide 10mg once weekly). The anticipated time on study treatment is 1 year, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-80 years of age;
* drug naive patients with type 2 diabetes uncontrolled with diet and exercise;
* tested negative for anti-glutamic acid decarboxylase (anti-GAD) antibodies;
* C-peptide (fasting) >=1.0ng/mL
* HbA1c >=6.5% and <=10.0% at screening;
* BMI >=25 (>23 for Asians) and <=45kg/m2 at screening;
* stable weight +/- 5% for at least 12 weeks prior to screening.

Exclusion Criteria:

* history of type 1 diabetes mellitus or acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma in the previous 6 months;
* evidence of clinically significant diabetic complications;
* symptomatic poorly controlled diabetes;
* myocardial infarction, coronary artery bypass surgery, post-transplantation cardiomyopathy or stroke within the previous 6 months;
* known hemoglobinopathy or chronic anemia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Safety: Adverse events, vital signs, physical examination, clinical laboratory tests, ECG and anti-taspoglutide antibodies. | Throughout study
Change from baseline in fasting plasma glucose; change from baseline in body weight. | 24 weeks
Responder rates for HbA1c (target <=7.0%, <=6.5%); relative change in glucose, insulin, C-peptide and glucagon during a meal tolerance test; beta cell function. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- United States (10):
  - Phoenix, Arizona
  - Los Angeles, California
  - Santa Ana, California
  - Avon, Indiana
  - Pahrump, Nevada
  - Charlotte, North Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - San Antonio, Texas
  - Richmond, Virginia
- Australia (2):
  - Adelaide
  - St Leonards
- Guatemala City, Guatemala
- Israel (6):
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Tel Aviv
- Mexico (6):
  - Acapulco
  - Aguascalientes
  - Chihuahua City
  - Hermosillo
  - Mexico City
  - Morelia
- Peru (2):
  - Lima
  - San Isidro
- Romania (5):
  - Bucharest
  - Buzău
  - Cluj-Napoca
  - Ploieşti
  - Tg. Mures
- Russia (7):
  - Chelyabinsk
  - Jaloslave
  - Moscow
  - S. Petersburg
  - S.petersburg
  - Saint Petersburg
  - Yaroslavl
- Slovakia (5):
  - Dolný Kubín
  - Levice
  - Prešov
  - Trenčín
  - Žilina
- Taiwan (4):
  - Changhua
  - Tainan
  - Taipei
  - Tapei County
- Ukraine (3):
  - Chernivtsi
  - Kiev
  - Lviv